CLINICAL TRIAL: NCT00787163
Title: Open Randomized Trial Comparing Perinatal Outcome Following Expectant Management Versus Amnioinfusion in PPROM <25 Wks With Persistent Oligohydramnios
Brief Title: Amnioinfusion Initiative
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Brescia (Other)
Collaborators: KU Leuven (Other); University of Milan (Other); Catholic University, Italy (Other)
Responsible Party: Anna Locatelli, University of Milano Bicocca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Amnioinfusion-001
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2008-11

CONDITIONS: Oligohydramnios
Keywords: pPROM; oligohydramnios; amnioinfusion; prematurity; Early premature rupture of membranes in pregnancy
MeSH Terms: conditions — Oligohydramnios; Preterm Premature Rupture of the Membranes; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): amnioinfusion
  Interventions: Procedure: amnioinfusion
- 2 (No Intervention): expectant management

INTERVENTIONS:
Procedure: amnioinfusion — serial amnioinfusions aimed at restoring amniotic fluid volume
  Arms: 1

SUMMARY:
The aim of this study is to compare perinatal survival in patients presenting with early spontaneous PPROM and persistent oligohydramnios, managed either conservatively or with serial amnioinfusions.

DETAILED DESCRIPTION:
Early spontaneous Preterm Premature Rupture of Membranes (PPROM) is associated with high perinatal mortality. Due to pulmonary hypoplasia and preterm delivery, mortality exceeds 60% when PPROM occurs prior to 24 weeks. When oligohydramnios persists, it may raise to 90%. Morbidity in survivors is also significant. In uncontrolled series, serial amnioinfusions, which have acceptable invasiveness and are of limited complexity, mortality was reduced to 60%.

We propose an open, multicenter randomized trial comparing perinatal survival in patients presenting with early spontaneous PPROM and persistent oligohydramnios, managed either conservatively or with serial amnioinfusions. Inclusion criteria: Single pregnancy, early spontaneous PPROM < 24.3 weeks, oligohydramnios (deepest vertical pocket < 2 cm) for at least 4 days and no longer than 15 days at enrolment. The study is open and will be run through a dedicated password protected web site, and with a minimal number of outcome measures. Primary outcome: Survival till discharge from the NICU. Secondary outcomes: Latency time from PPROM to delivery, gestational age at birth, indication for delivery, number of days of ventilatory support, serious neurologic morbidity, neonatal sepsis prevalence, need for oxygen at 36 weeks post-conception.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years, who are able to consent, with
2. Singleton pregnancy
3. with a normal structural examination as much as possible;
4. At least 2 US examination after pPROM for gestational age confirmation and diagnosis of persistent oligohydramnios
5. Follow up ultrasound examinations weekly in the treatment group
6. Acceptance of randomisation and to comply with the protocol

Exclusion Criteria:

1. Maternal contra-indications to intervention or prolongation of pregnancy, including severe medical conditions in pregnancy that make fetal intervention riskful;
2. Preterm labour defined as contractions >6/hour associated with cervical changes, cervix shortened (<15 mm at randomization),
3. Cervical cerclage in place
4. Chorioamnionitis, defined as 2 or more of the following: maternal temperature>38 degrees, foul-smelling vaginal discharge, uterine tenderness, fetal tachycardia>170 bpm, white blood cell count >18,000
5. Fetal structural anomaly detected at prenatal ultrasonography, or fetal chromosomal abnormalities involving autosomes
6. Previous invasive procedure in this index pregnancy
7. Fetal condition mandating immediate delivery
8. Severe bleeding
9. Maternal HIV and HCV infection
10. Multiple gestation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Survival of neonates/infants at discharge after serial amnioinfusions compared to survival after expectant management | discharge of every neonate from NICU

SECONDARY OUTCOMES:
Gestational age of delivery (main secondary outcome) | time of delivery for every case

CONTACTS AND LOCATIONS:
Overall Officials: Anna Locatelli, MD, Principal Investigator — University of Milano Bicocca; Patrizia Vergani, MD, Study Chair — University of Milano Bicocca
Locations (1):
- University of Milano Bicocca, Ospedale san Gerardo Monza, Monza, Milano, Italy